CLINICAL TRIAL: NCT06508606
Title: A Phase II Study of AK117 (Anti-CD47) Combined With Anti-EGFR in the Treatment of Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: AK117 (Anti-CD47) + Anti-EGFR for R/M HNSCC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Lei Liu, professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20241106
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — dexamethasone-(C21-phosphoramide)-(anti-EGFR)

STUDY DESIGN:
Intervention Model Description: A single-arm Phase II clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD47 (AK117) + anti-EGFR (Experimental): Patients meeting the inclusion criteria were given AK117 45mg/kg (D1, IVGTT, Q3W) in combination with anti-EGFR (initial dose 400mg/m2, subsequent doses of 250mg/m2, D1, QW) maintained for one year or until progression or intolerable toxicity occurred
  Interventions: Drug: AK117; Drug: anti-EGFR

INTERVENTIONS:
Drug: AK117 — AK117: 45mg/kg (D1, IVGTT, Q3W maintained for one year or until progression or intolerable toxicity occurred
Drug: anti-EGFR — anti-EGFR:initial dose 400mg/m2, subsequent doses of 250mg/m2, D1, QW) maintained for one year or until progression or intolerable toxicity occurred

SUMMARY:
The administration of first-line pembrolizumab monotherapy or combined chemotherapy has been shown to improve survival among patients with recurrent or metastatic head and neck squamous cell carcinoma (R/M HNSCC). However, over 80% of the patients still experience disease progression within a year. Upon progression, treatment options are notably constrained, typically comprising methotrexate, docetaxel, and cetuximab. The median progression-free survivaland overall survival following chemotherapy, targeted therapy, or their combination are dismally low, ranging from 2-3 months and 6-8 months, respectively. The clinical trials CheckMate 141 and KEYNOTE 040 have led to the approval of Nivolumab and Pembrolizumab as second-line treatments for R/M HNSCC. Nevertheless, the response rates to immune monotherapy are limited, ranging from 10% to 35%. Even after receiving standard second-line immunotherapy, over 80% of patients encounter disease progression within 6 months, and more than 60% succumb to the disease within a year. Therefore, there is a dearth of a standardized treatment for R/M HNSCC after the failure of first- or second-line PD-1 (L1) inhibitors and/or platinum-based therapy

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically or cytologically confirmed R/M HNSCC (including oral, oropharyngeal, hypopharyngeal, and laryngeal sites); Recurrence that cannot be cured by local treatment, and previous treatment with PD-1 (L1) inhibitors and/or platinum-based chemotherapy has failed.
2. At least one measurable lesion according to RECIST v1.1, excluding previously irradiated lesions unless clear progression occurred more than 3 months after the last radiotherapy;
3. Known HPV p16 status of oropharyngeal cancer;
4. Known PD-L1 expression status;
5. ECOG performance status of 0-1;
6. Expected survival ≥ 3 months;
7. Adequate bone marrow function, defined as: Hb ≥ 9.0 g/dL (90 g/L); ANC ≥ 1,500/mcL (1.5 × 10^9/L); PLT ≥ 100,000/mcL (100 × 10^9/L) and no blood transfusion within 3 weeks or growth factor (G-CSF, EPO) therapy within 2 weeks prior to dosing;
8. Adequate liver function, defined as: TBIL ≤ 1.5× upper limit of normal (ULN); If no liver metastases, AST and ALT ≤ 2.5× ULN; if liver metastases are present, AST or ALT ≤ 3.0× ULN; ALP ≤ 1.5× ULN; if liver metastases ≤ 2× ULN; Serum albumin ≥ 30g/L;
9. Adequate coagulation function: INR or PT, APTT ≤ 1.5× ULN. Participants on anticoagulant therapy should have these laboratory indices closely monitored;
10. Adequate renal function, defined as creatinine ≤ 1.5× ULN or Ccr ≥ 50 mL/min calculated using the Cockcroft-Gault formula corrected for body surface area;
11. Baseline left ventricular ejection fraction (LVEF) ≥ 50% measured by multiple-gated acquisition (MUGA) or echocardiogram (ECHO);
12. No severe organic heart disease or arrhythmias;
13. Women of childbearing potential (aged 15-49 years) must have a negative pregnancy test within 7 days before starting treatment. Both male and female participants of reproductive potential must agree to use effective contraceptive measures during the study period and for 3 months after discontinuation of treatment;
14. Voluntary signed informed consent by the study participant.

Exclusion Criteria:

1. Participants who have received treatment with cetuximab in the first line.
2. Grade ≥2 peripheral neuropathy (according to CTCAE 5.0).
3. Anticipated need for surgery or any other form of systemic or local anti-tumor therapy during the study, including maintenance therapy or radiotherapy for head and neck squamous cell carcinoma (excluding palliative treatment for non-target lesions).
4. Received systemic chemotherapy within 3 weeks prior to first administration of study drug, received small molecule targeted therapy within 2 weeks prior to first administration or within 5 half-lives (whichever is longer), received anti-tumor biologic therapy, large molecule targeted therapy or immunotherapy within 4 weeks prior to first administration, or underwent major surgery (excluding minor surgery within 2 weeks with complete recovery); received radiotherapy within 14 days prior to first administration of study drug (excluding central nervous system radiotherapy which requires a washout period of ≥28 days).
5. Known active central nervous system metastases and/or carcinomatous meningitis. Participants with treated brain metastases may participate if stable, without progressive or new neurological deficits, seizures, evidence of increased intracranial pressure, vomiting, or headaches.
6. Lesions that are superficially ulcerated or have broken through at baseline.
7. Residual toxicity from prior anti-tumor therapy (excluding alopecia, fatigue, and grade 2 hypothyroidism) or clinically significant laboratory abnormalities > grade 1 (CTCAE v5.0).
8. Pulmonary embolism or deep vein thrombosis within 3 months prior to first administration of study drug.
9. Known history of malignant tumors.
10. Any severe or uncontrolled systemic disease, including poorly controlled hypertension, diabetes.
11. History of active bleeding, coagulation disorder, or participants receiving coumarin anticoagulant therapy.
12. Known active hepatitis B or hepatitis C. Active hepatitis B is defined as known HBsAg positive and HBV DNA ≥500 IU/mL.
13. Concurrent severe, uncontrolled infections or known human immunodeficiency virus (HIV) (HIV antibody positive) infection, or diagnosis of acquired immune deficiency syndrome (AIDS); or poorly controlled autoimmune disease; or history of allogeneic tissue/organ transplant, stem cell or bone marrow transplant, or prior solid organ transplant.
14. Active bacterial, viral, fungal, rickettsial, or parasitic infections requiring systemic anti-infective therapy (unless treated and resolved before administration of study drug).
15. Received live virus vaccination within 30 days prior to first administration of study drug. Use of inactivated seasonal influenza vaccine or approved COVID-19 vaccine is allowed, with a washout period of >1 week prior to first administration of study drug.
16. History of or concurrent interstitial pneumonia, severe chronic obstructive pulmonary disease with respiratory failure, severe pulmonary insufficiency, symptomatic bronchospasm.
17. Received immunological therapy for any reason, including long-term use equivalent to >10 mg/day prednisone within 7 days prior to first administration of study drug or at any time during the study.
18. Uncontrolled pleural, peritoneal, pelvic effusion, or pericardial effusion requiring drainage ≥1 time per month.
19. Pregnancy test positive or breastfeeding participants. Women and men participants who do not plan to take adequate contraceptive measures within 180 days after the end of treatment.
20. Any other disease or clinically significant laboratory parameter abnormalities, severe medical or psychiatric condition, including substance abuse including alcohol abuse, which the investigator believes may compromise the safety of the participant, the integrity of the study, participant's ability to participate in the study, or interfere with the study objectives and result analysis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Adverse Events (AEs) | Up to approximately 1 years
  Characterization of incidence, severity and abnormal clinically significant laboratory findings of AEs
OS | Up to approximately 1 years
  overall survival

SECONDARY OUTCOMES:
ORR | Up to approximately 1 years
  Objective response rate
PFS | Up to approximately 1 years
  Progression Free Survival
DCR | Up to approximately 1 years
  Disease control rate
DoR | Up to approximately 1 years
  Duration of Response